CLINICAL TRIAL: NCT07103109
Title: Impact of Proximal Motor Control Exercise on Scapular Muscles Activation Pattern Post Mastectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ahram Canadian University (Other)
Collaborators: Benha University (Other)
Responsible Party: Principal Investigator, Mahmoud H Mohamed, PhD, Associate Professor, Ahram Canadian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Scapular Ms -Mastectomy 2025
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-08

CONDITIONS: Post Mastectomy
Keywords: Proximal stabilization

STUDY DESIGN:
Intervention Model Description: This is a parallel group randomized controlled trial
Who Masked: Participant
Masking Description: This is a parallel group randomized controlled trial with two arms receiving different interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental)
  Interventions: Other: Proximal stabilization exercises; Other: Conventional physical therapy
- control (Active Comparator)
  Interventions: Other: Conventional physical therapy

INTERVENTIONS:
Other: Proximal stabilization exercises — Patients will receive Scapular mobilization in five manners, superior glide, inferior glide, up-ward rotation, down-ward rotation, and distraction. Each mobilization will be done ten times. A thirty second break will be given between each set. Also scapular strengthening exercises composed of diagonal two (D2) flexion pattern to augment the upper, middle, lower, and serratus anterior muscles' activity level. To activate upper trapezius muscle, shoulder shrug exercise will be used. To activate serratus anterior muscle, Wall slide exercise will be used. Scapular retraction exercise for rhomboids and middle trapezius activation will be done. Strengthening exercises will be performed using weights were initiated with two sets of ten repetitions, beginning with a weight of 0.5 kg and progressed to 0.75, and1kg, it will be applied 5 days per week for 6 weeks
  Arms: study group
Other: Conventional physical therapy — Patients will receive shoulder joint mobilization, posterior capsular stretching, and ROM exercises in form of Codman/pendulum exercise. To mobilize the shoulder joint, distraction of the glenohumeral joint, posterior glide and caudal glide will be performed to the patients in a supine lying position at a frequency of two to three oscillations/second for one to two minutes. Every direction was repeated three to four times. At the resting position rhythmic oscillations grade I and II will be applied. In posterior capsule stretching each stretch will be repeated ten times for 20 seconds, between each stretching a 30-second break will be given. Pendulum exercise will be demonstrated to the patient at first, then they will performed it in the forward-backward direction, side-to-side direction, and circular pattern, for two to three minutes in each direction, it will be applied 5 days per week for 6 weeks

SUMMARY:
Mastectomy after breast cancer is usually accompanied by shoulder dysfunction which interferes with the daily life activities of the patients and causes physical and psychological impairments.

This study aims to assess the impact of strength and stabilization exercise on scapular muscles activation pattern after mastectomy.

DETAILED DESCRIPTION:
A total of 80 patients (n=40 per group), aged 35-55 years, diagnosed with shoulder dysfunction post mastectomy will be recruited for this study. Participants will be recruited from Baheya Hospital and National Cancer Institute. Participants will be screened for eligibility prior to being enrolled in the study participating in the study assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Post-mastectomy female subjects.
2. Age between 35-55 years.
3. All patients have shoulder dysfunction (three months to four months post mastectomy).

Exclusion Criteria:

1. Participants who have rheumatoid arthritis.
2. History of trauma or injuries.
3. Neurological deficits (stroke, Parkinsonism).
4. History of surgery on involved shoulder.
5. Diabetic patient.
6. Patients who rejected to participate in the trial, or to summit the formal consent form.

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Post-mastectomy female subjects
Enrollment: 60 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2026-06-10 (Estimated); Study Completion 2026-08-10 (Estimated)

PRIMARY OUTCOMES:
EMG Muscle Activation Amplitude | Baseline and 6 weeks
  Surface electromyography (sEMG) will be used to assess the activation patterns of scapular and rotator cuff muscles during functional tasks, such as shoulder flexion, abduction, and external rotation. The sEMG assessment will be conducted using a wireless sEMG system with a sampling rate of 2000 Hz and a bandwidth of 20-500 Hz. Pre-gelled, disposable, self-adhesive Ag/AgCl electrodes will be placed on the muscle belly according to SENIAM guidelines, with an inter-electrode distance of 20 mm. (serratus anterior, upper and lower trapezius, supraspinatus, and infraspinatus) during functional tasks.

SECONDARY OUTCOMES:
Shoulder pain and disability index (SPADI) | Baseline and 6 weeks
  It is a self-administered questionnaire that was found to be both sensitive and reliable. It contains thirteen items, which assess two domains (pain and disability). The patient circled the best number that reflected their ache or impairment on a scale from 0 to 10, which has an 8- items subscale to evaluate disability and a fiveitems subscale to measure pain. To calculate a final percentage score for assessing shoulder dysfunction, the scores from the two aspects were averaged

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Naeem, Ph.D, Study Director — Faculty of Physical Therapy, Beni Sueif university
Locations (3):
- Egypt (3):
  - Out patient clinic , faculty of Physical Therapy, Ahram Canadian university, Giza, Giza Governorate
  - Out patient clinic , faculty of Physical Therapy, Benha university, Banhā, Qualiobia
  - Out patient clinic , faculty of Physical Therapy, Beni Sueif university, Banī Suwayf

IPD SHARING:
Plan to Share IPD: Undecided